CLINICAL TRIAL: NCT02668692
Title: Efficacy and Safety of LEO 80185 Gel (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Japanese Subjects With Psoriasis Vulgaris
Brief Title: LEO 80185 Gel (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Japanese Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0076-1128
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis Vulgaris
Keywords: LEO 80185 gel, calcipotriol, betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 80185 gel (Experimental)
  Interventions: Drug: LEO 80185 gel
- Dovobet ® ointment (Active Comparator)
  Interventions: Drug: Dovobet ® ointment

INTERVENTIONS:
Drug: LEO 80185 gel — calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g, applied once daily to psoriasis lesions
  Arms: LEO 80185 gel
Drug: Dovobet ® ointment — calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g, applied once daily to psoriasis lesions
  Arms: Dovobet ® ointment

SUMMARY:
To compare the efficacy and safety of LEO 80185 gel with Dovobet® ointment in the treatment of psoriasis in Japanese subjects.

DETAILED DESCRIPTION:
A phase 3, national, multi-centre, 4-week, prospective, randomised, controlled, parallel-group, open trial of LEO 80185 gel versus Dovobet® ointment in Japanese subjects with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent has been obtained.
* 2. Japanese subjects
* 3. Aged 20 years or above
* 4. Clinical diagnosis of psoriasis vulgaris amenable to topical treatment of less than or equal to 30% BSA
* 5. A target psoriasis lesion on the scalp and on the non-scalp area of the body, each lesion of a minimum size of 10 cm2 and scoring at least 2 (mild) for each of the clinical signs (redness, thickness and scaliness).
* 6. Females of childbearing potential must have a negative result for a urine pregnancy test at Day 1 (Visit 1) and must agree to use an adequate method of birth control.
* 7. Able to communicate with the (sub)investigator and understand and comply with the requirements of the trial.

Exclusion Criteria:

* 1. Systemic use of biological treatments with a potential effect on psoriasis vulgaris
* 2. Systemic treatments with all therapies other than biological treatments with a potential effect on psoriasis vulgaris
* 3. PUVA therapy, UVB therapy or UVA therapy
* 4. Topical treatment of psoriasis on the areas to be treated with trial medication
* 5. Topical treatment of psoriasis on the face, genitals or skin folds with vitamin D analogues, potent or very potent corticosteroids or immunosuppressants
* 6. Topical treatment of conditions other than psoriasis with vitamin D analogues, potent or very potent corticosteroids or immunosuppressants
* 7. Planned initiation of, or changes in, concomitant medication that may affect psoriasis vulgaris
* 8. Patients with any of the following disorders (a) or symptoms (b) present on the areas to be treated with trial medication: (a) viral (e.g., herpes or varicella) lesions of the skin, fungal, spirochetal or bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, atrophic skin, striae atrophicae, ichthyosis, acne rosacea, ulcers, burns, frostbite, wounds, animal skin disease (scabies, crabs, lice, etc.) or (b) fragility of skin veins.
* 9. Other inflammatory skin diseases that may confound the evaluation of psoriasis vulgaris.
* 10. Erythrodermic, exfoliative or pustular psoriasis
* 11. Planned excessive exposure of areas to be treated with trial medication to either natural or artificial sunlight
* 12. Known or suspected disorders of calcium metabolism associated with hypercalcaemia, or albumin-corrected serum calcium above the reference range
* 13. Known or suspected severe renal insufficiency, severe hepatic disorders or severe heart disease.
* 14. Known or suspected hypersensitivity to any components of the investigational products.
* 15. Clinical signs or symptoms of Cushing's disease or Addison's disease
* 16. Treatment with any non-marketed drug substance
* 17. Current participation in any other interventional clinical trial
* 18. Previously randomised in this trial
* 19. Females who are pregnant, wishing to become pregnant or are breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Medical Corporation Bikyukai Kokubu Dermatology, Kitami-shi, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial had 213 participants enrolled and 206 participants randomized.
Groups:
- Dovobet® Ointment: Dovobet® ointment: calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g, applied once daily to psoriasis lesions
Period: Overall Study
Arm/Group | LEO 80185 Gel | Dovobet® Ointment
Started | 101 | 105
Completed | 100 | 105
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 80185 Gel | Dovobet® Ointment | Total
Number analyzed (Participants) | 101 | 105 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (13.7) | 54.3 (14.2) | 52.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 84 | 151
  Male | 34 | 21 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 101 | 105 | 206

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 'Overall Improvement' for the Target Lesion on the Scalp
Description: 'Overall improvement' for the target lesion on the scalp, defined as 'substantial resolution' of clinical signs and/or at least 'moderately improved' in the general change in the lesion.
  'Substantial resolution' is defined as a clinical score for thickness and scaliness of 0 and a clinical score for redness of 1 or less in the severity of clinical signs of the lesion.
Time Frame: End of Week 4
Population: All 206 randomised subjects are included in the full analysis set (FAS): 101 in the LEO 80185 group and 105 in the Dovobet® group.
  The per protocol analysis set (PPAS) was defined by excluding subjects from the FAS based on a review of protocol deviations. PPAS includes 94 subjects in the LEO 80185 group and 100 in the Dovobet® group.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel | Dovobet® Ointment
Number analyzed (Participants) | 101 | 105
Participants
  Overall improvement | 99 | 101
  Not overall improvement | 2 | 4
Statistical Analysis 1: Comparison: LEO 80185 Gel vs Dovobet® Ointment; Statistical analysis of the FAS; Test type: Superiority; p = 0.68, Fisher Exact; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.35 to 10.95]
Statistical Analysis 2: Comparison: LEO 80185 Gel vs Dovobet® Ointment; Statistical analysis of the PPAS; Test type: Superiority; p = 0.68, Fisher Exact — Treatment comparison by Fisher's exact test; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.34 to 10.72] — Odds of 'overall improvement' in LEO 80185 gel group relative to Dovobet® ointment group

2. Secondary Outcome: Number of Subjects With 'Overall Improvement' for the Target Lesion on the Non-scalp Area of the Body
Description: 'Overall Improvement' for the target lesion on the non-scalp area of the body, defined as 'substantial resolution' of clinical signs and/or at least 'moderately improved' in the general change in the lesion.
  'Substantial resolution' is defined as a clinical score for thickness and scaliness of 0 and a clinical score for redness of 1 or less in the severity of clinical signs of the lesion.
Time Frame: End of Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel | Dovobet® Ointment
Number analyzed (Participants) | 101 | 105
Participants
  Overall improvement | 83 | 99
  Not overall improvement | 18 | 6
Statistical Analysis 1: Comparison: LEO 80185 Gel vs Dovobet® Ointment; Statistical analysis for the FAS; Test type: Superiority; p = 0.009, Fisher Exact; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.11 to 0.74]
Statistical Analysis 2: Comparison: LEO 80185 Gel vs Dovobet® Ointment; Statistical analysis of the PPAS; Test type: Superiority; p = 0.003, Fisher Exact — Treatment comparison by Fisher's exact test; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.08 to 0.63] — Odds of 'overall improvement' in LEO 80185 gel group relative to Dovobet® ointment group

3. Secondary Outcome: The Change in the Sum of the Scores (Total Sign Score) for the Severity of the 3 Clinical Signs:Thickness, Scaliness, Redness From Baseline to End of Week 4 (Visit 1-4) for Each Target Lesion.
Description: Severity was recorded for each of the 3 clinical signs according to the 9-point scales* below.
  *intermediate intervals (0.5, 1.5, 2.5, 3.5) serve as mid points between the defined grades.
  Redness 0=none (no erythema)
  1. slight (faint erythema, pink to very light red)
  2. mild (definite light red erythema)
  3. moderate (dark red erythema)
  4. severe (very dark red erythema)
  Thickness 0=none (no plaque elevation)
  1. slight (slight, barely perceptible elevation)
  2. mild (definite elevation but not thick)
  3. moderate (definite elevation, thick plaque with sharp edge)
  4. severe (very thick plaque with sharp edge)
  Scaliness 0=none (no scaling)
  1. slight (sparse, fine scale, lesions only partially covered)
  2. mild (coarser scales, most of lesions covered)
  3. moderate (entire lesion covered with coarse scales)
  4. severe (very thick coarse scales, possibly fissured)
  Negative change denotes a decrease in the score and therefore a decrease in disease severity.
Time Frame: From Baseline to end of Week 4 (Visit 1-4)
Population: The per protocol analysis set (PPAS) was defined by excluding subjects from the full analysis set (FAS) based on a review of protocol deviations. PPAS includes 94 subjects in the LEO 80185 group and 100 in the Dovobet® group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LEO 80185 Gel | Dovobet® Ointment
Number analyzed (Participants) | 94 | 100
Scores on a scale
  Scalp (PPAS) | -6.43 (1.91) | -6.79 (1.90)
  Non-scalp (PPAS) | -5.31 (2.44) | -6.46 (2.05)

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form up to 14 days after last visit (Week 4).
Arm/Group | LEO 80185 Gel | Dovobet® Ointment
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/105
Serious Adverse Events (participants affected / at risk) | 1/101 | 0/105
Other Adverse Events (participants affected / at risk) | 13/101 | 9/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 80185 Gel (N=101) | Dovobet® Ointment (N=105)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 80185 Gel (N=101) | Dovobet® Ointment (N=105)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Chelitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Kaposi's varicelliform eruption (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days